CLINICAL TRIAL: NCT04972877
Title: Effect of Electro-acupuncture on Ovarian Function and Outcome of IVF-ET of Women With Diminished Ovarian Reserve：a Randomized Controlled Clinical Trial
Brief Title: Effect of Electro-acupuncture on Women With Diminished Ovarian Reserve
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Huazhong University of Science and Technology (Other)
Collaborators: Wuhan No.1 Hospital (Other); Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other); The Affiliated Hospital of Jiangxi University of Traditional Chinese Medicine (Other); Edwatz Medical Research Institude (Unknown); Wuhan Jinxin Gynecology and Obstetrics Hospital of Integrative Medicine (Unknown)
Responsible Party: Principal Investigator, Dongmei Huang, Department of Integrated Traditional Chinese and Western Medicine Tongji hospital Affiliation: Huazhong University of Science and Technology, Huazhong University of Science and Technology
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TJ-IRB20190620
Record Dates: First submitted 2021-06-24; First posted 2021-07-22 (Actual); Last update posted 2021-07-22 (Actual); Status verified 2021-07

CONDITIONS: Diminished Ovarian Reserve
Keywords: Electro-acupuncture; Diminished ovarian reserve; In vitro fertilization-embryo transfer; Randomized controlled trial

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group (Active Comparator): Treatment group protocol：participants will receive electro-acupuncture twice or three times a week with a maximum of 24 times in 2-3 months. Each treatment session lasts for 30 minutes.
  Interventions: Other: Treatment group protocol
- Control group (Sham Comparator): Control group protocol：participants will receive sham electro-acupuncture twice or three times a week with a maximum of 24 times in 2-3 months. Each treatment session lasts for 30 minutes.
  Interventions: Other: Control group protocol

INTERVENTIONS:
Other: Treatment group protocol — For treatment group, two groups of acupoints will be used alternatively. The first group consists of some acupoints. The patients will be asked to stay in supine position. Disposable sterilized needles (Size: 0.25*40/50 mm) will be inserted into a depth of 15~35 mm and stimulated manually to evoke needle sensation. And then some acupoints will be thereafter connected to electrical stimulators and stimulated with low-frequency and the maximum tolerated intensity of the patients. The other needles without electrical stimulators will be manually stimulated to evoke "Deqi" every 10 minutes.
  The second group consists of other acupoints. Patients will be asked to stay in prone position. The stimulation will be in the same way as the first group.
  Arms: Treatment group
Other: Control group protocol — For control group, four pseudo-acupoints are used, with two points on each shoulder and the two on each upper arm, which are not located on any meridians. The patients will be asked to stay in supine position and keep the whole body relaxed and comfortable. Disposable sterilized needles (Size: 0.18*25 mm) will be inserted superficially to a depth of < 5 mm without any manual stimulus and the needle sensation ("Deqi" in TCM) should not be evoked. Electrodes are connected to the needles, but the stimulators should be turned on at an intensity of zero. Each intervention lasts for 30 minutes.
  Arms: Control group

SUMMARY:
Diminished ovarian reserve (DOR) is the precursor state of ovarian failure, and can cause the decline of women's reproductive function. Some studies have demonstrated that acupuncture can improve ovarian function. In this trial, we hypothesize that electro-acupuncture is efficient for the ovarian function and the following outcome of IVF-ET in DOR patients.

DETAILED DESCRIPTION:
First, patients will be recruited according to the inclusion criteria and exclusion criteria.

Second, baseline measurements (including ovarian reserve function, blood biochemical index, scores from the self-rating anxiety and depression scale, quality of life) will be taken.

Third, each patient will receive 24 sessions of acupuncture in 2-3 months, twice or three times a week.

Last, the above baseline measurements will be taken again as soon as the treatment is finished and outcome measures will be recorded after the treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Age < 40, will undergo IVF-ET;
2. Low ovarian reserve: Antral follicle count (AFC)<7, or AMH<1.1ng/ml; or has a history of poor ovarian response: in the last hyper stimulation cycle, the number of retrieved oocytes<3;
3. Spouse' semen examination is normal, or after semen prewash can reach the standard of common IVF or Intracytoplasmic Sperm Injection(ICSI).

Exclusion Criteria:

1. Male with azoospermia;
2. Male/female's chromosome is abnormal;
3. Adenomyosis, uterine fibroids, endometrial polyps, scar uterine, reproductive system tuberculosis, oviduct effusion, pelvic lesions such as ovarian endometriosis cyst or tumor;
4. Female has other endocrine disease: thyroid diseases, hyperprolactinemia, insulin resistance, diabetes, adrenal diseases, etc.
5. Definitively diagnosed autoimmune diseases such as systemic lupus erythematosus, rheumatoid arthritis, antiphospholipid syndrome;
6. Other pathogenesis that leads to recurrent miscarriage or agnogenic recurrent miscarriage;
7. A history of cancer and has received radiotherapy and chemotherapy;
8. Had acupuncture treatment in recent 3 months;
9. Unwilling to sign the informed consent of this study.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 338 (Estimated)
Dates: Start 2019-09-09 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Assessing the change of ovarian reserve function | 0 week and up to 4 weeks
  Assessing patients' ovarian reserve function before and after electro-acupuncture intervention, including: (1) The serum AMH, inhibin, and FSH and E2 levels on the third day of menstruation;(2) AFC.

SECONDARY OUTCOMES:
Clinical pregnancy rate | through study completion, an average of 1 year
  the clinical pregnancy rate per cycle of IVF-ET after electro-acupuncture.
Outcomes of IVF | through study completion, an average of 1 year
  1. Gn dosage(U/d) and usage days;
  2. E2 level(pg/ml) and endometrial thickness(mm) on human chorionic gonadotropin (HCG) day;
  3. number of oocytes;
  4. MII oocytes;
  5. normal fertility rate;
  6. the number of available embryos;
  7. number of high-quality embryos;
  8. cycle cancellation rate (including cycle cancellation rate caused by various reasons);
  9. implantation rate: including fresh periodic implantation rate, per cycle implantation rate and cumulative implantation rate;
  10. fresh cycle clinical pregnancy rate and cycle cumulative clinical pregnancy rate;
  11. early, mid and late pregnancy abortion rate;
  12. risk of ovarian hypertrophy and incidence of obstetric complications;
  13. FSH(mIU/ml), LH(mIU/ml), E2(pg/ml) and AMH(ng/ml) in follicular fluid; Oxidative stress related indicators such as reactive oxygen species (ROS), superoxide dismutase (SOD) level, etc.;
  14. live rate: including fresh cycle live rate, cycle live rate and cumulative live rate.
Blood biochemical index examination | 0 week and up to 12 weeks
  Testing the levels of blood corticotrophin-releasing hormone (CRH), norepinephrine, adrenaline, 5-hydroxytryptamine, beta-aminobutyric acid (GABA), dopamine (DA) and neuro-endorphin of the patients before and after treatment.
Questionnaires | 0 week and up to 4 weeks
  Evaluation of anxiety, depression, quality of life and sleep state is performed before and after treatment.
  1. Baker anxiety self-rating scale (BAI) and baker depression self-rating scale (BDI-Ⅱ) : higher score indicates higher degree of depression or anxiety [12-13].
  2. Zung anxiety self-rating scale (Zung-SAS), Zung depression self-rating scale (Zung-SDS) [14-15].
  3. Quality of life measurement (QOL): Quality of life will be assessed by SF-36 and Chinese quality of life scale (CHQOL).
  4. Self-Rating Scale of Sleep (SRSS), sleep dysfunction rating scale (SDRS), Pittsburgh sleep quality index (PSQI).
Follow-up detection | through study completion, an average of 1 year
  Pregnancy patients will be followed up to the end of pregnancy. Adverse pregnancy outcomes and live birth rates will be recorded. Non-pregnant patients will be followed up for 1 year after treatment, testing the ovarian reserve function, follow-up treatment and pregnancy status of the patients within 1 year.

CONTACTS AND LOCATIONS:
Overall Officials: Dongmei Huang, doctor, Principal Investigator — Department of Integrated Traditional Chinese and Western Medicine Tongji hospital of Huazhong University of Science and Technology
Locations (1):
- Department of Integrated Traditional Chinese and Western Medicine Tongji hospital of Huazhong University of Science and Technology, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: Yes
we use the Clinical Trial Management Public Platform to manage and share our date.
Supporting Information: CSR
Time Frame: January, 2026, for 1 year
Access Criteria: only for research